CLINICAL TRIAL: NCT06305325
Title: eHealth Antenatal Coparenting Intervention to Prevent Postpartum Depression Among Primiparous Women, Karachi, Pakistan: A Pilot Randomized Controlled Trial
Brief Title: Coparenting Intervention to Prevent Postpartum Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brock University (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Salima Sulaiman, Assistant Professor, Brock University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 35957
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Postpartum Depression; Anxiety
Keywords: online; postpartum depression; Coparenting relationship
MeSH Terms: conditions — Depression, Postpartum; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: coparenting framework: it has 3 levels. First is the individual level, which consists of the parent's individual characteristics, which comprises of attitudes, parental beliefs, and emotional and mental health. It has a bidirectional relationship with coparenting and the overall inter-parental relationship. Individual child factors, such as temperament may also play a role in shaping the coparenting relationship. The second level is the family level. It comprises the overall interpersonal relationship, referring to the existing ability of couples to demonstrate support and respect for each other. It could influence the coparental relationship or in reverse, the coparental relationship may influence the overall inter-parental relationship. The third level is the extra-familial level. It has two components: support and stress that are based on a stress-coping perspective. The role of environmental support is viewed as enhancing the coparenting relationship
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): control group received the standard care. It included antenatal classes offered at the CC clinic, which comprised of four face-to-face sessions in clinic. These classes focus on pregnancy and postpartum care including baby growth in each trimester, minor discomforts, diet, exercise, personal hygiene, complications during pregnancy, labour and delivery stages, breastfeeding, care of newborn baby, and family planning methods. The 2-3 hour long face-to-face classes are offered every week on Saturdays in the clinic
- eHealth antenatal Coparenting Intervention (Experimental): This intervention focuses on developing conflict management, problem solving, communication, and mutual support to foster positive joint parenting of an infant. A modification in the delivery of this intervention was made in the current study in order to make it deliver online. The eACoP intervention included eight antenatal videos from Feinberg's Family Foundation intervention. A website for the eACoP intervention was developed, and all the videos were uploaded to the website. These videos were 30-40 minutes each. The videos were in English and subtitles in Urdu were added to the videos. These videos were accompanied by an activity-based coparenting workbook. The coparenting workbook includes a worksheet and homework for each video and was also translated into Urdu
  Interventions: Behavioral: eHealth Antenatal Coparenting Intervention

INTERVENTIONS:
Behavioral: eHealth Antenatal Coparenting Intervention — This intervention focuses on developing conflict management, problem solving, communication, and mutual support to foster positive joint parenting of an infant. A modification in the delivery of this intervention was made in the current study in order to make it deliver online. The eACoP intervention included eight antenatal videos from Feinberg's Family Foundation intervention. A website for the eACoP intervention was developed, and all the videos were uploaded to the website. These videos were 30-40 minutes each. The videos were in English and subtitles in Urdu were added to the videos. These videos were accompanied by an activity-based coparenting workbook. The coparenting workbook includes a worksheet and homework for each video and was also translated into Urdu
  Arms: eHealth antenatal Coparenting Intervention

SUMMARY:
The goal of this pilot randomized controlled trial was to examine the feasibility and acceptability of an ehealth antenatal coparenting intervention (eACoP) in primiparous Pakistani women. The secondary purpose of the study was to see the effectives of the intervention in prevention postpartum depression in women. Two hundred and twelve primiparous couples were randomized into an intervention or a control group from the Aga Khan University Hospital. Couples were randomized using consecutively numbered sealed envelopes. Couples in the intervention group received the eACoP intervention during pregnancy, consist of eight online videos in addition to the standard care provided at the center. Both the intervention group and control group received standard care.

ELIGIBILITY:
Inclusion Criteria:

* primiparous
* Both women and their partners willing to participate and indicated by signed consent
* Up to 24 weeks of gestation (first and second trimester of pregnancy)
* Singleton pregnancy
* Able to speak, read, and understand English or Urdu
* Have access to internet

Exclusion Criteria:

* Did not have access to internet
* Had an EPDS score of >12.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-09-23 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2020-02-22 (Actual)

PRIMARY OUTCOMES:
feasibility-recruitment rate, adherence, and follow-up rate | recruitment-at the time of recruitment during pregnancy pre intervention, adherence rate-during the intervention, follow up rate- 6 weeks and 12 weeks after the delivery of an infant
  feasibility refers to how well the eACoP intervention was implemented. It included recruitment rate, adherence, and follow-up rate. The recruitment log was completed to assess the recruitment rate by the Research Assistant (RA) at the time of recruitment and used to determine a) eligibility rate; b) enrollment rate; c) refusal rates; and d) reasons for non-participation. The eligibility rate was defined as the percentage of screened people who met eligibility criteria. The enrollment rate was defined as the percentage of eligible couples who consented to take part in the study. The intervention Activity Log was completed by the RA weekly by telephone to assess the adherence rate and used to determine a) compliance with intervention material and reasons for non-compliance; and b) completion of workbook and reasons for not completion. The non-compliance form was used to assess reasons for non-compliance. The follow-up rate recorded on follow-up log
Acceptability- Participants satisfaction | immediately after the intervention
  It is a 14-item self-report questionnaire designed to measure an individual's satisfaction with an intervention which also included four open ended questions. Higher scores indicate higher levels of satisfaction.

SECONDARY OUTCOMES:
Depressive Symptoms | baseline, 4-6 weeks and 12-weeks postpartum
  Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self-report measure, asking about the depressive symptomatology during the past week. It is a reliable and valid instrument with a sensitivity of 85% and specificity of 77%. The sensitivity of the Urdu version is 98%. Each item is scored on a four-point scale with a total score ranges from 0-30. The minimum is 0 and the maximum total score is 30. Couples who score greater than twelve are likely to be suffering from depressive symptomatology.
anxiety | baseline, 4-6 weeks and 12-weeks postpartum
  The State-Trait Anxiety Inventory (STAI) is a twenty item self-report questionnaire with each item scored on a four-point Likert scale; 1 = "not at all" to 4 = "very much so", with a total score ranging from 20 to 80. Couples who score > 40 are likely to be suffering symptoms of anxiety. Internal consistency of the STAI-S ranges from 0.91 to 0.95. The coefficient alpha of the Urdu version was 0.87.
Coparenting Relationship | baseline, 4-6 weeks and 12-weeks postpartum
  The Coparenting Relationship Scale (CRS) was used to measure coparental quality in couples. The CRS is a thirty-five item self-report questionnaire, consisting of seven subscales. It has good reliability and strong stability with Cronbach's alphas ranging from 0.91 to 0.94 across genders. Each item is scored on a seven-point Likert scale from "that is not true of us" (score 0) to "very true of us" (score 6). Six of the scales are scored on the same Likert scale except exposure to conflict scale which is scored on six-point Likert scale from "never" (score 0) to "several times a week" (score 6). The CRS tool is in English and was translated into Urdu. The Urdu version was back translated into English. the pilot testing of the tool was done with ten pregnant couples from a community Health Center (CHC), an out-patient clinic at the Aga Khan University Hospital (AKUH), were asked to complete the scale.
Relationship Satisfaction- couple relationship satisfaction to discriminate between distressed and non-distressed relationship. | baseline, 4-6 weeks and 12-weeks postpartum
  The Revised Dyadic Adjustment Scale (RDAS) was used to measure couple relationship satisfaction and discriminate between distressed and non-distressed relationship. The RDAS has 14 items, each of which asks the respondents to rate certain aspects of their relationship on a six-point Likert scale. Only one question "Do you and your mate engage in outside interests together"? ask the respondents to rate on a five-point Likert scale. Scores on the RDAS range from 0 to 69 with higher scores indicating greater relationship satisfaction and lower scores indicating greater relationship distress. The cut-off score for the RDAS was ≥ 48 such that scores of 48 and above indicate non-distress and scores of 47 and below indicates relationship distress. Cronbach's alpha for the RDAS is 0.90. The RDAS has been used in the postpartum population in previous studies.
Postpartum Childcare Stress | 12-weeks postpartum
  The Postpartum Childcare Stress Checklist (PCSC) was used to identify parental perceptions of childcare stress. The PCSC has 19 items, asking the participants to rate their experience of events mentioned in the items over the past 4 weeks. Each item is rated as "yes or (1)" or "No or (2)". The PCSC explores the participant's experience related to the relationship with the partner, caring for the infant, social interactions, and establishing a new routine. Scores on the PCSC range from 1 to 19 with higher scores indicating lower childcare stress and lower scores indicating greater childcare stress. The PCSC had internal consistency of 0.81 (Dennis et al., 2018). The PCSC tool is available in English and was translated into Urdu. The Urdu version was back translated into English. The tool has not been used in Pakistan and has not been tested for reliability and validity for this population
Infant Development | 12 weel postpartum
  The Ages and Stages Questionnaire (ASQ-3) was used to identify infants at risk of delays in development at communication, gross motor, fine motor, problem solving, and personal-social domains at 12-week postpartum. The ASQ-3 is comprised of 30 age-appropriate questions to which parents respond with three categories: yes (10 points), sometimes (5 points), and not yet (0 points). Scores for each area range from 0 to 60 with higher scores indicating lower risk of delays in overall development. It is a reliable and valid instrument with a sensitivity and specificity of 87.4% and 95.7% respectively
partner support | baseline and 12 weeks postpartum
  The Postpartum Partner Support Scale (PPSS) is a new instrument, which was used to measure postpartum partner support in couples. The PPSS tool is a twenty-item self-report, asking about the partner support during the past four weeks. Each item is scored on a four-point Likert scale; 1 = "Strongly Disagree" to 4 = "Strongly Agree. Higher scores are indicative of a more positive partner support. The Cronbach's alpha for the PPSS is 0.96. The PPSS tool is available in English and was translated into Urdu.

CONTACTS AND LOCATIONS:
Overall Officials: Salima Sulaiman, PhD, Principal Investigator — Brock University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
IPD are confidential and linked to participants ID. I am bound with Ethics Review to nor disclose their information

REFERENCES:
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Dennis CL, Brown HK, Brennenstuhl S. The Postpartum Partner Support Scale: Development, psychometric assessment, and predictive validity in a Canadian prospective cohort. Midwifery. 2017 Nov;54:18-24. doi: 10.1016/j.midw.2017.07.018. Epub 2017 Jul 29. PMID 28780475
- [Background] Dennis CL, Brown HK, Brennenstuhl S. Development, Psychometric Assessment, and Predictive Validity of the Postpartum Childcare Stress Checklist. Nurs Res. 2018 Nov/Dec;67(6):439-446. doi: 10.1097/NNR.0000000000000308. PMID 30067584
- [Background] Spielberger, C. D., Gorsuch, R. L., Lushene, R., Vagg, P. R., & Jacobs, G. A. (1983). Manual for the State-Trait Anxiety Inventory. Palo Alto, CA: Consulting Psychologists Press.
- [Background] Spanier, G. B. (1976). Measuring dyadic adjustment: New scales for assessing the quality of marriage and similar dyads. Journal of Marriage and the Family, 38(1), 15-28. https://doi.org/10.2307/350547
- [Background] Squires, J. & Bricker, D. (2009). Ages & Stages Questionnaires [R], (ASQ-3): A Parent- Completed Child-Monitoring System. Brookes Publishing Company.
- [Background] Feinberg ME, Brown LD, Kan ML. A Multi-Domain Self-Report Measure of Coparenting. Parent Sci Pract. 2012 Jan 1;12(1):1-21. doi: 10.1080/15295192.2012.638870. Epub 2012 Jan 20. PMID 23166477